CLINICAL TRIAL: NCT04103658
Title: Near-infrared Heating of Skin to Delineate Non-melanoma Skin Cancer Lesions: a Pilot Study.
Brief Title: NIR and Skin Cancer Margins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Kiersten Pianosi, MD, Western University, Canada
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114153
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Non-melanoma Skin Cancer

STUDY DESIGN:
Masking Description: Patients will be randomly assigned to the group of excision without or with near-infrared heat. Both the patient and investigator will be aware of the group allocation prior to the definitive excision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (control) (No Intervention): This will be the standard of care group. The excision of the non-melanoma skin cancer will be based on standard visual inspection with 4-6mm margins.
- NIR heating (Experimental): This will be the NIR heating group, where the excision of the non-melanoma skin cancer will be based on the lesion margins based on the application of near-infrared radiation (with 4-6mm margins).
  Interventions: Radiation: Near-infrared heating

INTERVENTIONS:
Radiation: Near-infrared heating — Same as the arm/group description. The NIR heating group will have the non-melanoma skin cancer lesion excised based on the lesion borders established from application of NIR heat at a distance of 20cm for 10 minutes.
  Arms: NIR heating

SUMMARY:
We aim to determine whether the application of near-infrared radiation via standard heat lamp to non-melanoma skin lesions (such as basal cell carcinomas) before surgical excision is able to better delineate the lesion and surgical margins. If found to do so, pre-heating of skin lesions could lead to more specimens with negative margins. Patients presenting to the tertiary care centre skin cancer clinic for excision of skin cancer will be approached and offered to participate in the study.

DETAILED DESCRIPTION:
Non-melanoma skin cancer (NMSC) is the most common cancer diagnosis in Canada, and its incidence is still increasing. Visual examination followed by biopsies of suspicious lesions are the gold standard for skin cancer diagnosis. The mainstays of treatment include photodynamic therapy, radiation therapy, and surgical excision. The margins of NMSC lesions are typically determined via visual inspection, and excised based on delineating normal from abnormal tissue. According to the National Comprehensive Cancer Network, low-risk basal cell cancers should be excised with a 4mm margin; squamous cell skin cancers and high-risk basal cell cancers should be excised with 4-6mm margins, as per the National Comprehensive Cancer Network. These lesions frequently occur on cosmetically sensitive areas of the head and neck, therefore accurate margins and excision can help to preserve the overall appearance. Accurate lesion delineation with proper margins can also reduce the need for further treatment if the margins are positive. In approximately 2-3% of cases at our centre, the margins are positive.

Near-infrared radiation (NIR) represents the light spectrum from 0.7 to 1.5 micrometers. At the shorter wavelengths, it merges with the red spectrum of visible light. These forms of light have the ability to heat the skin up to a 5 mm depth. Previous studies have examined the relationship between skin blood flow and temperature when heating skin, where dermal temperature can reach a certain peak in a defined time. Other studies have investigated the application of NIR when combined with photo immunotherapy, as a means of treating other cancers. More elaborate multispectral analysis devices have been studied for their effectiveness in diagnosing cutaneous malignancies. NIR application is well tolerated, in past studies.The objective of this study is to determine if the vasculature of normal skin and NMSC skin appears differently following heating with NIR light, and if this difference corresponds to better margin delineation.

The excisions and reconstructions are all within the standard of care. The only added testing will be application of near-infrared heat via a heating lamp to the lesional skin, for a total of ten minutes. Each patient will have their skin cancer lesion photographed, and traced onto acetate film. The NIR heating will then occur under a lamp for a total of ten minutes at a distance of 20cm. At the end of the ten minutes, the lesion and its borders will again be traced onto a separate acetate film. Using Excel for block randomization, patients will then be randomized to excision with the non-heated versus heated margins. The allocation will not be known until the moment of assignment. The excisions will then occur in the same fashion between the two groups, and all specimens will be submitted for pathology, as is standard of care.

Data will be recorded for various patient and lesions factors that may potentially influence the outcome of NIR heating therapy. These include age and gender, lesion size and location, and history of skin disorders. The lesion size and final pathology, with quantitative margin distances, will be recorded. Statistical analysis will be performed to determine if there is an overall difference in qualitative (negative or positive) and quantitative margin status between those lesions excised under standard procedure vs. NIR heating.

ELIGIBILITY:
Inclusion Criteria:

The patient population includes individuals with a nonmelanotic cervicofacial cutaneous malignancy referred to a tertiary care skin cancer clinic for definitive treatment. Patients must have:

* Histologically confirmed nonmelanotic cutaneous malignancies, either basal cell or squamous cell carcinoma
* No prior treatment with investigational agents
* Ability to tolerate intended treatment Patient's age is greater than or equal to 18 years

Exclusion Criteria:

* Prior radiation therapy or photodynamic therapy to the area with the NMSC lesion
* Patients with a history of cutaneous photosensitization
* Unable to consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Margin status | 3 months
  Difference in margin status between the control and the near-infrared heating group.

SECONDARY OUTCOMES:
Skin vascularity changes | 3 months
  Visual changes in the vasculature of normal skin and NMSC skin following application or NIR light.

IPD SHARING:
Plan to Share IPD: No